CLINICAL TRIAL: NCT02270918
Title: A Phase I Placebo-Controlled, Open-Label, Crossover Study to Assess the Reversibility of Apixaban Anticoagulation With the Four Factor Prothrombin Complex Concentrate Kcentra in Healthy Volunteers
Brief Title: Reversibility of Apixaban Anticoagulation With the Four Factor Prothrombin Complex Concentrate Kcentra
Acronym: 4PAR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Bristol-Myers Squibb (Industry); CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 14P.366
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Thrombosis
Keywords: Xa inhibitor; Prothrombin complex concentrate; anticoagulation
MeSH Terms: conditions — Thrombosis; Hemophilia B | interventions — apixaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apixaban with Kcentra (Active Comparator): Oral apixaban will be administered to steady state in healthy volunteers followed by a single infusion of prothrombin complex concentrate Kcentra at 25 units/Kg
  Interventions: Drug: Kcentra; Drug: Apixaban
- Apixaban with placebo (Placebo Comparator): Oral apixaban will be administered to steady state in healthy volunteers followed by a single infusion of saline
  Interventions: Drug: Apixaban; Drug: Placebo

INTERVENTIONS:
Drug: Kcentra — IV infusion
  Other Names: 4 factor prothrombin complex concentrate
  Arms: Apixaban with Kcentra
Drug: Apixaban
Drug: Placebo
  Arms: Apixaban with placebo

SUMMARY:
Apixaban is an anticoagulant (also known as blood thinner) approved by the Food and Drug Administration (FDA) for reducing the risk of stroke and systemic embolism in patients with non-valvular atrial fibrillation. It has no reliable method of reversal. Kcentra is an FDA approved drug derived from blood that is used as an antidote to treat people with bleeding associated with taking the well-known anticoagulant warfarin. This is a Phase I, placebo-controlled, single site, open-label, crossover trial to evaluate the reversibility apixaban anticoagulation with Kcentra.

DETAILED DESCRIPTION:
Oral anticoagulants are effective in the treatment and prevention of venous and arterial thrombotic events. For more than 50 years the only class of anticoagulant available had been the vitamin K antagonist (VKA), warfarin, which requires frequent blood work for monitoring. Apixaban is a new approved anticoagulant that is used to treat patients who have blood clots or are at risk for developing blood clots. Unlike warfarin, the use of apixaban does not require frequent blood work for monitoring and is associated with lower bleeding risk. All anticoagulation therapies are associated with spontaneous or provoked bleeding risk and reversal of their blood thinning effects might be needed. Reversal of anticoagulation may also be needed in cases where emergent or urgent surgery is indicated. There is currently no available reversal agent for apixaban. Prothrombin complex concentrate (PCC) contain clotting factors and can replace factors inhibited by anticoagulants. In a recent study in the Netherlands a four factor prothrombin complex concentrate, Cofact (not available in the USA) was shown to be able to reverse the anticoagulation effects of another factor Xa inhibitor, rivaroxaban. Kcentra is a four factor prothrombin complex concentrate that was FDA approved in 2013 and is used as an antidote to treat people with bleeding associated with taking warfarin. It contains clotting factors II, VII, IX and X derived from donated blood and could be effective in reversing the anticoagulation effects of the factor Xa inhibitor, apixaban. No effective reversal agent for apixaban exists. Physicians struggle with bleeding in patients who are on apixaban. Indeed, this is not an uncommon problem for patients who suffer brain bleeds or trauma. This study could potentially identify Kcentra as reversal agent for patients taking apixaban. This study will test the hypothesis that Kcentra has the potential to significantly reduce the anticoagulation effect of apixaban as measured by thrombin generation assay at 30 minutes post infusion of Kcentra as compared to placebo infusion in subjects dosed to steady state with apixaban.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible for participation in this trial, the subject must:

  1. Be a healthy male or female between ages 18-55 (inclusive) at the screening visit
  2. Have a body mass index (BMI) >19 and <33 (inclusive)
  3. If a female, subject

     1. Can be of childbearing potential and must demonstrate a urine β-hCG level consistent with the nongravid state at the pretrial (screening) visit and agree to use (and/or have their partner use) an acceptable method of birth control beginning at the pretrial visit throughout the trial (including washout intervals between treatment periods) and until 2 weeks after the last dose of trial drug in the last treatment period.
     2. Can be of non-childbearing potential which is defined as: a female who is postmenopausal without menses for at least 1 year and an Follicle stimulating hormone value in the postmenopausal range upon pretrial (screening) evaluation and/or a female who is status post hysterectomy, oophorectomy or tubal ligation
     3. Must be off hormonal oral or transdermal contraceptives for at least 4 weeks prior to initial dose of trial drug
  4. Be a nonsmoker for at least approximately 6 months
  5. Have serum creatinine level < 1.5 mg/dL
  6. Have a prothrombin time (PT) and activated partial thromboplastin time (PTT) level below the upper limit of normal
  7. Have platelet count within normal limits
  8. Be willing to refrain from the use of anticoagulants and antiplatelet medications including aspirin and non-steroidal anti-inflammatory drugs (NSAIDs) during the entire period of study participation
  9. Be willing to provide written informed consent for the trial
  10. Be willing to comply with trial restrictions

Exclusion Criteria:

1. Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological (including stroke and chronic seizures) abnormalities or diseases
2. Has history of cancer (excluding treated cutaneous squamous or basal cell carcinoma of >3 years previous)
3. Has history of venous or arterial thromboembolic disease
4. Has a history of clinically significant bleeding risks including prior serious head trauma
5. Has had major surgery within 6 months prior to screening visit
6. Is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies for 2 weeks prior to trial start date until the post-trial visit
7. Is unable to refrain from using any drugs or substance known to be inhibitors or inducers of cytochrome P450 (CYP) enzymes including grapefruit products for 2 weeks prior to dosing and throughout the study, until the post-trial visit
8. Has a history of illicit drug abuse within six months prior to screening visit
9. Consumes greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce]) per day and cannot refrain from alcohol for the duration of the trial
10. Has a history of significant multiple and/or severe allergies (e.g. food, drug), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
11. Has known anaphylactic or severe systemic reactions to any components of study drugs (including heparin induced thrombocytopenia) or contraindication to the administration of PCC or any other related blood products.
12. Has moderate or severe hepatic disease or other clinically relevant bleeding risk
13. Has positive history for hepatitis B surface antigen, hepatitis C or HIV
14. Has first degree relatives with history of bleeding disorder or hypercoagulable disease
15. Use of any drugs or products which at the discretion of the investigator would increase bleeding risk
16. Is considered inappropriate for participation by the investigator for any reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
thrombin generation assay (TGA) | 30 minutes

SECONDARY OUTCOMES:
Anti-factor Xa activity | 30 minutes

OTHER OUTCOMES:
prothrombin time (PT) | 30 minutes
activated partial thromboplastin time (PTT) | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Walter K Kraft, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hosptial, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Nagalla S, Thomson L, Oppong Y, Bachman B, Chervoneva I, Kraft WK. Reversibility of Apixaban Anticoagulation with a Four-Factor Prothrombin Complex Concentrate in Healthy Volunteers. Clin Transl Sci. 2016 Jun;9(3):176-80. doi: 10.1111/cts.12398. Epub 2016 May 12. PMID 27170068